CLINICAL TRIAL: NCT04324697
Title: Evaluation of Anterior Alveolar Ridge Reconstruction With Allogenic Bone Plate and Autogenous Cortical Bone Chips: A Radiographic and Histological Clinical Study
Brief Title: Radiographic and Histological Evaluation of Regenerated Bone After Grafting Using Allograft Shell and Autogenous Chips
Acronym: Shell grafting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: October 6 University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Khalid Tarek Mohamed Karkar, Teaching assistant, October 6 University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS-2018-03M
Record Dates: First submitted 2020-03-23; First posted 2020-03-27 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-04

CONDITIONS: Alveolar Bone Resorption
Keywords: Allograft; Autogenous chips; Horizontal augmentation; Khoury shell technique

STUDY DESIGN:
Intervention Model Description: Reconstruction of the localized deficient anterior maxilla using an allograft cortical bone plate, which was fixed at a distance from the alveolar ridge using two micro-screws, and the created gap between the allograft plate and the alveolar ridge was filled with autogenous cortical bone chips harvested intraorally using a bone scrapper.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Horizontal alveolar bone augmentation — Horizontal augmentation in anterior maxilla using allograft shell and autogenous chips with no need for a second surgical site
  Other Names: MAXGRAFT@Cortico - Botiss

SUMMARY:
The clinical cases in the present study described the khoury shell technique using an allograft plate and autogenous chips, for horizontal reconstruction of the anterior alveolar ridge in the esthetic zone. Without need to use autogenous bone graft techniques that are characterized by more aggressive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with class IV of Cawood and Howell classification in the anterior maxilla.
* Males and females 18-50 years of age.
* Patients with adequate oral hygiene.
* Patients with healed sites for at least 6 months after tooth extraction.
* Patients with an inter-arch distance of at least 6 mm.
* Compliance with all requirements in the study and signing the informed consent.

Exclusion Criteria:

* Patients with diseases of the immune system or systemic disease affecting bone healing
* Patients who are chronic users of medications known to affect the periodontal status.
* Patients with history of intravenous and/or oral bisphosphonate use.
* Pathologic lesions or acute infection in the area of defect.
* Patients who are pregnant or lactating mothers.
* Heavy smokers who smoke more than 10 cigarettes a day.
* Patients with poor oral hygiene that are not amenable to motivation and improvement.
* Patients with history of irradiation of the head and neck region.
* Vulnerable patients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Alveolar Bone quantity | 6 months
  Alveolar bone width by millimeters using Cone Beam Computed Tomography

SECONDARY OUTCOMES:
Alveolar Bone quality | 7 months
  Histological evaluation of status of regenerated bone vitality and remodeling

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No